CLINICAL TRIAL: NCT01874418
Title: Study for Usefulness and Standardization of CSF and Blood Biomarkers in Alzheimer's Disease
Brief Title: Biomarker Study to Diagnose Alzheimer's Disease
Acronym: ADAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, SangYun Kim, Department of Neurology, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ADAM
Record Dates: First submitted 2013-06-03; First posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biomarker study (Other): Oligomeric beta-amyloid 42 in serum, as well as, monomeric beta-amyloid 42, total tau and phosphorylated tau in CSF
  Interventions: Other: Biomarker

INTERVENTIONS:
Other: Biomarker — Oligomeric beta-amyloid 42 in serum, as well as, monomeric beta-amyloid 42, total tau and phosphorylated tau in CSF

SUMMARY:
The purpose of our study is to investigate CSF and blood biomarkers among the subjects with mild cognitive impairment (MCI) and Alzheimer's disease (AD) as well as normal controls.

DETAILED DESCRIPTION:
Alzheimer's disease is the most prevalent cause of dementia. A biomarker is a variable that are measured in vivo and indicate specific features of disease related molecular mechanisms and pathologic changes, including amyloid processing and aggregation, tau hyperphosphorylation, accumulation of neurofibrillary tangles, synaptic dysfunction, neurodegeneration, and loss of brain tissue.

We examine serum oligomeric beta-amyloid 42 and CSF monomeric beta-amyloid 42, total tau and phosphorylated tau, as well as PiB-PET, FDG-PET and brain MRI in 90 participants (30 normal controls, 30 patients with mild cognitive impairment, 30 patients with Alzheimer's disease).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent obtained from the subject or the subject's legally acceptable representative ( if applicable) in accordance with the local regularities.
2. Both male and female, aged > 50 and <90, if women, must have no childbearing potential
3. Controls did not have subjective memory complaints or any of 28 diseases and did not have a history suggestive of a decrease in cognitive function (stroke or transient ischemic attack, seizures, Parkinson's disease, multiple sclerosis, cerebral palsy, Huntington's disease, encephalitis, meningitis, brain surgery, vascular surgery of the brain, diabetes requiring insulin control, improperly managed hypertension, cancer diagnosed within the past 3 years excluding skin cancer, shortness of breath while sitting still, use of home oxygen, heart attack with changes in memory, walking, or solving problems lasting at least 24 hours afterwards, kidney dialysis, liver disease, hospitalization for mental or emotional problems in the past 5 years, current use of medications for mental or emotional problems, alcohol consumption greater than 3 drinks each day, drug abuse in the past 5 years, treatment for alcohol abuse in the past 5 years, unconsciousness for more than one hour other than during surgery, overnight hospitalization due to head injury, illness causing a permanent decrease in memory or other mental functions, trouble with vision that prevents reading ordinary print even with glasses, or difficulty understanding conversations because of hearing even with a hearing aid)
4. The controls also had scores that were at least one standard deviation above the mean scores of the respective age- and education-matched population on the K-MMSE and an average score of 0.42 or less on the Korean Instrumental Activities of Daily Living (K-IADL)

Exclusion Criteria:

-

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Oligomeric beta-amyloid 42 in serum | baseline
  To compare oligomeric beta-amyloid 42 in serum among normal controls, MCI and AD

SECONDARY OUTCOMES:
Total tau concentration in CSF | baseline
  To compare total tau concentration in CSF among normal controls, MCI and AD
Phosphorylated tau concentration in CSF | baseline
  To compare phosphorylated tau concentration in CSF among normal controls, MCI and AD
Monomeric beta-amyloid 42 in CSF | baseline
  To compare monomeric beta-amyloid 42 in CSF among normal controls, MCI and AD

OTHER OUTCOMES:
PiB PET | baseline
  To compare the uptake of PiB PET among normal controls, MCI and AD
FDG-PET | baseline
  To compare the pattern of hypometabolism with FDG-PET among normal controls, MCI and AD
Brain MRI | baseline
  To compare the volumetry and surface morphometry of brain T1-weighted MRI among normal controls, MCI and AD

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea